CLINICAL TRIAL: NCT07365839
Title: CLeAR: Pilot Study to Evaluate the Efficacy of Cemiplimab (PD-1 Inhibition) With or Without Fianlimab (LAG-3 Inhibition) After Y90 Radioembolization in Patients With Hepatocellular Carcinoma
Brief Title: Cemiplimab +/- Fianlimab Post Y90 Radioembolization in Patients With Hepatocellular Carcinoma
Acronym: CLeAR
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-24-21103
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Treatment with cemiplimab (Experimental): 350 mg cemiplimab intravenous (IV) every 3 weeks
  Interventions: Drug: Arm 1 cemiplimab
- Arm 2 Treatment with (Experimental): 350 mg cemiplimab intravenous (IV) + 1600 mg fianlimab intravenous (IV) every 3 weeks
  Interventions: Drug: Arm 2 cemiplimab and fianlimab

INTERVENTIONS:
Drug: Arm 1 cemiplimab — Cemiplimab 350mg IV every 3 weeks up to 1 year.
  Other Names: Libtayo, Anti-PD-1 antibody
  Arms: Arm 1 Treatment with cemiplimab
Drug: Arm 2 cemiplimab and fianlimab — Cemiplimab 350mg IV and fianlimab 1600mg every 3 weeks up to 1 year
  Other Names: Libtayo, Anti-PD-1 antibody & Anti-LAG-3 antibody
  Arms: Arm 2 Treatment with

SUMMARY:
Randomized, 2-arm, non-comparative, pilot study assessing the efficacy of cemiplimab with or without fianlimab after treatment with yttrium-90 (Y90).

DETAILED DESCRIPTION:
At 2-8 weeks after yttrium-90 (Y90) radioembolization, patients will be randomized to receive treatment with cemiplimab or with a fixed-dose combination of cemiplimab and fianlimab. If Y90 is administered in 2 treatments, the first dose of the study treatment must be given no more than 12 weeks after first Y90 treatment and at least 2 weeks after the second treatment. Patients will receive the assigned study treatment once per 3-week cycle and will continue treatment for up to 17 cycles (approximately 1 year) or until disease progression or intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma (HCC) in the liver by radiographic imaging or histology
* Eligible for yttrium-90 (Y90) treatment by the following definition:

Patients must have lung dose threshold for Y90 glass microspheres of 30 Gy (≤ 30 Gy per treatment for glass) and an estimated future liver remnant volume (FLRV) ≥ 30% of whole liver volume

* Age ≥18 years
* Disease in the liver measurable by modified Response Evaluation Criteria in Solid Tumors (mRECIST)
* Child Pugh Scale Score A-B7
* Not eligible for (according to the practice of the treating institution) or declined the following treatments:

  * surgical resection
  * immediate liver transplantation
  * thermal ablation
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Troponin (TnT and TnI) ≤1 × upper limit of normal (ULN) at baseline Note: Patients with TnT or TnI levels between >1 to 2 × ULN are permitted if repeat levels within 24 hours are ≤1 × ULN. If TnT or TnI levels are >1 to 2 × ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on the medical judgement in the patient's best interest.
* Alkaline phosphatase ≤5 × ULN
* Aspartate aminotransferase (AST) ≤5 × ULN
* Alanine transaminase (ALT) ≤5 × ULN
* Creatinine clearance >30 mL/min (actual or calculated per the Cockcroft-Gault formula)
* Bilirubin ≤2 milligram/ deciliter (mg/dL) Exception: If a patient has documented Gilbert's syndrome and a total bilirubin is ≥2 mg/dL, the total bilirubin requirement may be waived provided the direct bilirubin is within normal limits (WNL)
* Patients with known Human immunodeficiency virus (HIV) infection are eligible if the following conditions are met:

  * the HIV is well controlled with no AIDS-related complications
  * undetectable viral load
  * Cluster of Differentiation 4 (CD4)+ T-lymphocyte count(T-cell) above 350 cells/microliters (μL) Note: HIV testing is not required for study participation.
* Patients with known active hepatitis B virus (HBV) infection are eligible if the following conditions are met:

  * serum HBV Deoxyribonucleic Acid (DNA) polymerase chain reaction ( PCR)below the limit of detection
  * receiving anti-HBV treatment Note: HBV testing for diagnosis is not required for study entry. Determination of known active HBV infection is based on medical history.
* Patients with known chronic hepatitis C virus (HCV) infection are eligible if they have undetectable HCV RNA by PCR Note: HCV testing for diagnosis is not required for study entry. Determination of known chronic HCV infection is based on medical history. Receipt of anti-HCV medication has no bearing on study eligibility.
* Patients with HIV or hepatitis must have established longitudinal care with a qualified specialist (eg, infectious disease or hepatologist).

Note: at the time of enrollment, the specialist providing longitudinal care must be documented in the source medical record.

- Women of childbearing potential (WOCBP) must have a negative serum beta-Human Chorionic Gonadotropin (hCG) at screening WOCBP are defined as women who are fertile following menarche until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high Follicle-Stimulating Hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the Clinical Trials Facilitation Group (CTFG) guidance20.

- WOCBP are required to practice highly effective contraception during the entire trial and for at least 6 months after the last dose of study treatment. Highly effective contraceptive measures include the following:

* Stable use of combined (estrogen and progestogen containing) hormonal contraception or progestogen-only hormonal contraception (oral, injectable, or implantable) associated with inhibition of ovulation initiated 8 weeks before the screening serum beta-hCG test
* Intrauterine device (IUD); intrauterine hormone-releasing system (IUS)
* Vasectomized partner, provided that the male vasectomized partner is the sole male sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure
* Sexual abstinence, defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs, if evaluated by the treating investigator to be reliable in relation to the duration of required contraception (up to 18 months) and the preferred and usual lifestyle of the participant.

Note: period abstinence (calendar, symptothermal, post-ovulation methods), withdrawal, spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.

* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire trial and for at least 6 months after the last dose of study treatment
* Male study participants with WOCBP partners are required to use condoms during the entire trial and for at least 6 months after the last dose of study treatment unless they are vasectomized or practice sexual abstinence.

  * Vasectomized study participants must have received medical assessment of surgical success for the procedure.
  * Sexual abstinence, defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs, must be evaluated by the treating investigator to be reliable in relation to the duration of required contraception (up to 18 months) and the preferred and usual lifestyle of the participant.
* Male study participants must agree not to donate sperm during the entire trial and for at least 6 months after the last dose of study treatment

Exclusion Criteria:

* Any history of invasive malignancy within the past 3 years, except for the following:

  * adequately treated basal cell or squamous cell skin cancer, localized prostate cancer, breast ductal carcinoma in situ, low-grade endometrial carcinoma, or in situ cervical cancer,
  * localized prostate cancer under active surveillance or gonadotropin-releasing hormone (GNRH) therapy
  * treating physician determines previous cancer has been adequately treated with high probability for cure (as documented in medical record)
* Presence of extrahepatic disease Note: non measurable (<1 centimeter (cm)) lesions outside the liver are acceptable if they do not represent a deterrent for Y90 treatment per the standards of the treating institution
* Receipt of more than 1 prior embolization (TACE or Y90) treatment/procedure
* Portal vein thrombosis (PVT) Vp3 or Vp4
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (except viral hepatitis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or myocarditis
* Current enrollment in any other investigational therapeutic drug study
* Currently breastfeeding
* Recipient of an organ transplant, including bone marrow allogeneic transplant
* Previous systemic therapy for HCC
* Ongoing or recent (within 2 years) autoimmune disorder except for the following:

  * Vitiligo
  * Alopecia
  * Hashimoto's thyroiditis
  * Celiac disease controlled by diet
  * Chronic skin conditions that do not require systemic therapy
  * Childhood asthma that has resolved
  * Residual hypothyroidism that requires only hormone replacement
* Use of immunosuppressive medication within 14 days before the first dose of study treatment, except the following:

  * include topical, inhaled, local injection or intranasal steroids
  * systemic steroids at doses of ≤10 mg/day of prednisone (equivalent)
  * steroids for premedication
* TnT or troponin I TnI ≥ 2 × ULN at baseline
* History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (eg, cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks before the first dose of study treatment
* Active infection requiring treatment (except HIV/hepatitis as noted in inclusion criteria)
* Diagnosis of immunodeficiency that is related to, or results in, chronic infection (except HIV/hepatitis as noted in inclusion criteria) or is related to organ or allogeneic bone marrow transplant
* Known hypersensitivity to the active substances or to any of the excipient
* Received a live vaccine within 30 days before the planned start of study medication. Note that this applies to live or live attenuated vaccination with replicating potential
* Prior history of interstitial lung disease or pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2035-02-28 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of cemiplimab with or without fianlimab as measured by progression-free survival (PFS) | Baseline, 6, 12, and 18 months, then every 6 months until off study up to 5 years
  Progression-free survival, defined as the number of days from the start date of Y90 treatment (administered two times) to the date of progression, relapse, or death.

SECONDARY OUTCOMES:
Evaluate the safety and toxicity profile of cemiplimab with or without fianlimab based on the number of patients experiencing grade greater than grade 3 treatment-related adverse events (TRAE). | Baseline through 90 days following end of treatment (EOT) up to 5 years
  Incidence of treatment-related grade ≥3 adverse events as defined in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0). Adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans.
Assess the objective response rate (ORR) for patients receiving cemiplimab with or without fianlimab. | 6, 12, and 18 months
  The percentage of patients who have a complete response (CR) and a partial response (PR) as measured by Modified (Response Evaluation Criteria in Solid Tumors) (mRECIST). mRECIST is a method to adapt the RECIST 1.1 criteria to measure HCC specifically. mRECIST only takes the viable tumor into account, which allows necrosis of the tumor to not be mistaken for progression.
Assess the progression free survival (PFS) rate for patients receiving cemiplimab with or without fianlimab | 6, 12, and 18 months, then every 6 months until off study up to 5 years
  Using response from mRECIST criteria to determine date of progression for calculation of PFS
Assess the median overall survival (OS) for patients receiving cemiplimab with or without fianlimab. | 6, 12 and 18 months then every 6 months until off study up to 5 years
  Overall survival, defined as time from the date of Y90 treatment to the date of death by any cause, measured by the number of participants alive through study completion.
Assess the overall survival (OS) rate for patients receiving cemiplimab with or without fianlimab. | 6, 12 and 18 months, then every 6 months until off study up to 5 years
  Overall survival, defined as time from the date of Y90 treatment to the date of death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kinsey, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) at this time.